CLINICAL TRIAL: NCT05074719
Title: Characterization of the Index Individual for Contact Participants Enrolled in Clinical Trials of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Prevention Interventions; COVID-19 Prevention Trials Network (CoVPN) 3502-01
Brief Title: Index Individuals in SARS-CoV-2 Prevention Research Studies (COVID-19 Index Individuals Companion Study)
Acronym: IICov19PRS
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Fred Hutchinson Cancer Center (Other)
Responsible Party: Principal Investigator, Ruanne Barnabas, Associate Professor, School of Medicine: Global Health, University of Washington
Other Study IDs: STUDY00011462; 38771 (Registry Identifier: DAIDS, NIAID, NIH); 3502-01 (Other Grant/Funding Number: COVID-19 Prevention Network (CoVPN)); 3UM1AI068614-14S1 (NIH)
Record Dates: First submitted 2021-10-08; First posted 2021-10-12 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: SARS-CoV-2 Infection; COVID-19; Coronavirus Infection; SARS (Severe Acute Respiratory Syndrome)
Keywords: index; cofactors; transmission; prevention; mitigation; viral load; subgenomic RNA; exposure; long COVID; PASC (post-acute sequelae of SARS-CoV-2)
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Severe Acute Respiratory Syndrome; Erythema Multiforme; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1) mid-turbinate nasal swab sample and 2) dried blood spot sample (optional)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Cohort A comprises individuals that enroll within two weeks of diagnosis of SARS-CoV-2 infection. These individuals will be asked to provide a baseline mid-turbinate nasal swab for SARS-CoV-2 testing and complete questionnaires at baseline and on Days 7 and 14. Through these questionnaires, index individuals will report on the clinical course of their illness and share information about their household environment, including potential exposures there-in and any COVID-19 transmission mitigation strategies implemented (whether intentional or as part of standard home routines). Enrolled Cohort A index individuals will also be invited to participate in the SARS-CoV-2 Antibody Sub-study and provide a dried blood spot specimen (at baseline) for antibody testing.
- Cohort B: Cohort B comprises individuals that enroll more than two weeks after diagnosis of SARS-CoV-2 infection. These individuals will be asked to provide a mid-turbinate nasal swab for SARS-CoV-2 testing and to complete a questionnaire reporting retrospectively on their COVID-19 illness and household environment. Through this questionnaire, index individuals will report on the clinical course of their illness and share information about their household environment, including potential exposures there-in and any COVID-19 transmission mitigation strategies implemented (whether intentional or as part of standard home routines). These individuals will also complete a questionnaire reporting on the persistence and/or delayed onset of symptoms and complications that they associate with their COVID-19 illness. Enrolled Cohort B index individuals will also be invited to participate in the SARS-CoV-2 Antibody Sub-study and provide a dried blood spot specimen (at baseline) for antibody testing.

SUMMARY:
Clinical trials of prevention modalities for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection and coronavirus disease (COVID-19) and pneumonia are underway under separate protocol(s) for close contacts (i.e., household contacts, [e.g.,3502]) of infectious (index) individuals (3502-01).

Characterizing the index individuals within households will ascertain the risk of exposure for the contact participant. These data will be used to strengthen the precision of efficacy estimates.

This ancillary observational study will assess the cofactors for infectiousness among index individuals whose close contacts are enrolled in COVID-19 prevention clinical trials.

Additionally, this study will assess post-acute sequelae of SARS-CoV-2 infection in index individuals that are more than two weeks past their initial diagnosis.

DETAILED DESCRIPTION:
Within households, the incidence of SARS-CoV-2 is high, but the risk of transmission is characterized by exposure cofactors and transmission mitigation strategies.

Exposure cofactors are defined as cofactors that influence infectiousness of the index individual such as SARS-CoV-2 viral load, SARS-CoV-2 antibodies, and viable virus (as characterized by subgenomic RNA).

Transmission mitigation strategies are defined as modifiable cofactors that influence transmission and currently include physical distancing, social isolation, ventilation, and handwashing.

The continued progression of the pandemic has seen an increase in reports of persistent and/or delayed onset of symptoms and complications in patients well past the acute phase of COVID-19 infection. The prevalence and impacts of these post-acute sequelae of SARS-CoV-2 infection (PASC), which may continue for weeks to months after the initial COVID-19 illness, are not well understood.

Up to approximately 2,000 eligible index individuals who have close contacts (e.g., uninfected household members) in COVID-19 prevention research studies will be invited to participate. Individuals that enroll within two weeks of their diagnosis will be asked to provide a baseline mid-turbinate nasal swab for SARS-CoV-2 testing and complete questionnaires at baseline and on Days 7 and 14. Through these questionnaires, index individuals will report on the clinical course of their illness and share information about their household environment, including potential exposures there-in and any COVID-19 transmission mitigation strategies implemented (whether intentional or as part of standard home routines). Individuals that enroll more than two weeks after being diagnosed will be asked to provide a mid-turbinate nasal swab for SARS-CoV-2 testing and to complete a questionnaire reporting retrospectively on their COVID-19 illness and household environment. These individuals will also complete a questionnaire reporting on the persistence and/or delayed onset of symptoms and complications that they associate with their COVID-19 illness. Enrolled index individuals will also be invited to participate in the SARS-CoV-2 Antibody Sub-study and provide a dried blood spot specimen (at baseline) for antibody testing.

Working closely with prevention research studies, we propose to characterize the index individual level cofactors for SARS-CoV-2 transmission.

Each contact between an index individual and close contact is the unit of analysis for the research study.

The ascertainment of SARS-CoV-2 status among contacts/household members will be done through the parent prevention research study, e.g., through an existing clinical trials agreement with the CoVPN 3502/R 10933-10987-COV-2069 study.h

Across these studies, the investigators aim to assess:

* Prevalence and incidence of SARS-CoV-2 infection in the close contacts.
* Reported SARS-CoV-2 transmission mitigation strategies and exposures as assessed in the index individuals (3502-01) and household contact protocols (e.g., 3502) and the correlation between them.
* Association between the index individual SARS-CoV-2 viral load and subgenomic RNA and infection in the contact participant.
* Association of the duration of symptomatic COVID-19 in the index individual on the risk of SARS-CoV-2 transmission.
* Association of SARS-CoV-2 viral genotype in index individual to related SARS-CoV-2 genotype infection in the contact participant
* Post-acute sequelae of SARS-CoV-2 (PASC) infection in individuals that are weeks to months past their initial SARS-CoV-2 infection.

With these combined household data, effective, modifiable cofactors for household transmission can be identified to inform future post-exposure interventions. With the inclusion of data related to viral and host exposure cofactors, the investigators can increase the precision of predictive models of SARS-CoV-2 infection, adjusted for exposure and mitigation strategies. Data collected on PASC will contribute to the characterization of the long term consequences of SARS-CoV-2 infection and Post-acute COVID-19 Syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 and older; children and adolescents 10 years of age and older, at the time of signing the informed assent with parent or guardian consent
2. Willing and able to provide informed consent/assent with parental consent
3. Diagnosis of SARS-CoV-2 infection using a diagnostic test with a positive result, e.g., RT-PCR, antigen test, or other test format (approved or with Emergency Use Authorization issued by the US FDA or by local health authority) and within the eligibility period of the contact's prevention research study, or is currently being assessed for COVID-19
4. A close contact is being screened for enrollment or has enrolled in a SARS-CoV-2 prevention research study
5. Access to a smart phone or device with internet access to complete a questionnaire or communicate with research study team

Exclusion Criteria:

1. Hospitalization (current)
2. No household member enrolling/enrolled in a SARS-CoV-2 prevention research study

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is enrolling children and adolescents 10 years of age and older and adults 18 and older, identified as the index case(s) of SARS-CoV-2 infection within their households.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Prevalence and incidence of SARS-CoV-2 infection in the household contacts of index individuals | Day 1/Baseline for index individuals (3502-01); assessed weekly across 4 weeks for household contacts (3502)
  Positive SARS-CoV-2 reverse transcription-polymerase chain reaction (RT-PCR) test, or equivalent, as assessed in the Index Individuals Companion Study (3502-01) and household contact COVID-19 Prevention Study (3502) protocols
Characterization of reported SARS-CoV-2 transmission mitigation strategies | Across 14 days (Day 1/Baseline and Days 7 &14 Questionnaires) for index individuals, or retrospectively for individuals enrolled more than two weeks after diagnosis (3502-01); assessed at baseline and at 4 weeks for household contacts (3502)
  Characterization and quantification of reported SARS-CoV-2 transmission mitigation strategies as assessed in the index individuals (3502-01) and household contacts (3502) protocols. Assessment of concordance and/or correlation between index individuals' reporting and household contacts' reporting.
Assessment of household exposures | Across 14 days (Day 1/Baseline and Days 7 &14 Questionnaires) for index individuals, or retrospectively for individuals enrolled more than two weeks after diagnosis (3502-01); assessed at baseline and at 4 weeks for household contacts (3502)
  Characterization and quantification of household exposures assessed in the index individuals (3502-01) and household contacts (3502) protocols. Assessment of concordance and/or correlation between index individuals' reporting and household contacts' reporting.

SECONDARY OUTCOMES:
SARS-CoV-2 viral load and/or subgenomic RNA | Day 1/Baseline sample (single day) for index individuals (3502-01)
  SARS-CoV-2 semiquantitative RT-PCR and subgenomic RNA from the index individuals' mid-turbinate nasal swab (3502-01)
SARS-CoV-2 genotyping within households | Day 1/Baseline sample (single day) for index individuals; assessed weekly for household contacts, across 4 weeks.
  SARS-CoV-2 genotyping from a subset of index individuals' (3502-01) and household contacts' (3502) mid-turbinate nasal swab samples. Where feasible (per genotype sample availability), genotype comparisons among index and newly infected household (i.e. contacts) members.

OTHER OUTCOMES:
Serum-based antibodies to SARS-CoV-2 | An optional, Day 1/Baseline sample (single day) for index individuals (3502-01).
  Measurement of antibodies to SARS-CoV-2 in index individuals (3502-01) and household contacts (3502) based on dried blood spot sample(s).

CONTACTS AND LOCATIONS:
Overall Officials: Ruanne Barnabas, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington International Clinical Research Center, Seattle, Washington, United States